CLINICAL TRIAL: NCT05490940
Title: A Prospective Randomized Study to Evaluate Sensory Recovery of Digital Nerves After Primary Repair Performed by Microsurgical Epineural End-to-end Neurorrhaphy Alone, or in Combination With an Enwrapping With Fibrin Sealant Tisseel®
Brief Title: Sensory Recovery of Digital Nerves After Microsurgical Epineural Neurorrhaphy Alone or in Combination With Tisseel - RET
Acronym: RET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-02050
Record Dates: First submitted 2022-07-06; First posted 2022-08-08 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Digital Nerve Injuries
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, investigator-blinded, monocentric study
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is examiner- and patient blinded. While the operating surgeon is not blinded, postoperative examinations will be performed by physicians who do not know the group assignment of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microsurgical end-to-end neurorrhaphy alone (No Intervention): This group of patients receives a simple, tension-free, end-to-end microsurgical neurorrhaphy alone (without fibrin glue)
- Microsurgical end-to-end neurorrhaphy in combination with an enwrapping with fibrin sealant Tisseel® (Experimental): This group of patients receives a simple, tension-free, end-to-end microsurgical neurorrhaphy in combination with an enwrapping with fibrin sealant Tisseel®.
  Interventions: Drug: Tisseel®

INTERVENTIONS:
Drug: Tisseel® — The investigational medical product (IMP) in this study is Tisseel®, which is a tissue sealer consisting of two components:
  1. Sealer protein: Human fibrinogen as "glue" component and synthetic Aprotinin, which delays fibrinolysis.
  2. Human thrombin: Thrombin is an unique molecule that functions both as a procoagulant and anticoagulant. It activates platelets through its receptor on the platelets and regulates its own. generation by activating coagulation factors V, VIII and even XI resulting in a burst of thrombin formation.
  Its indications are a better hemostasis, enforcement of vessel/gastrointestinal sutures and tissue sutures (mesh grafts, flaps etc).
  Other Names: Neurorraphy alone
  Arms: Microsurgical end-to-end neurorrhaphy in combination with an enwrapping with fibrin sealant Tisseel®

SUMMARY:
Evaluation of sensitivity after primary surgical treatment of digital nerve injuries with microsurgical epineural end-to-end neurorrhaphy alone or in combination with the fibrin glue Tisseel®

DETAILED DESCRIPTION:
Lacerations of the fingers with nerve injuries are a common reason for a presentation at the surgical emergency ward of the Inselspital Bern. The patient complains of either reduced sensitivity or even complete numbness in the affected finger. This leads to a clear functional loss in daily activities and should be reliably tested during the clinical examination. If a nerve lesion is suspected, the wound and the affected nerve should be explored in the operating room. If the suspicion is confirmed, the sheath of the two nerve endings can be sewn under the microscope or with surgical loupes.

Tension free microsurgical epineural end-to-end neurorrhaphy of digital nerves after sharp or blunt lesions is a simple and effective procedure in order to regain sensory recovery and prevent neuroma formation.

Industry is promoting different aids in order to achieve better outcomes after repair - such as tissue glue, grafts and conduits. These products are more or less expensive, which becomes more and more important as the general cost in the Swiss health system are progressively increasing.

The aim of this randomized, prospective controlled study is thus to compare the clinical benefit of a primary epineural end-to-end neurorrhaphy combined with fibrin glue (Tisseel®) versus a simple epineural end-to-end neurorrhaphy alone.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Acute digital nerve lesion(s) distal to the superficial arterial arch on one or more fingers that qualify for primary direct end-to-end microsurgical epineural neurorrhaphy
* Age ≥18 years

Exclusion Criteria:

* Lesions that do not allow a tension-free direct suture, partial transections, amputation, re-vascularisation
* Age < 18 years
* Pre-operation on the injured finger
* Clinical comparison with contralateral finger not possible (e.g. due to amputation).
* Treatment that is known to inhibit the growth/regeneration of nerves impaired or can cause neuropathy - such as chemo- or radiotherapy before or during the whole study
* Systemic and local neurological impairments (polyneuropathy, diabetes mellitus, carpal tunnel syndrome, etc.)
* History of vascular diseases like Raynaud's disease syndrome that affects blood flow or sensation in the upper can affect the extremities
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, or dementia
* Women who are pregnant (urin pregnancy test) or breast feeding. Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Contraindications to the investigational product, e.g. known allergy to components of the Tisseel® fibrin glue
* Participation in another interventional study within the 30 days preceding and during the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
two point discrimination | preoperative
  For this purpose a standardized two-point-discriminator (PADGETT DeMayo Two-Point Discrimination Device, Used for Post hand surgery diagnostic. MFID: PM-855) is used
two point discrimination | 6 weeks postoperative
  For this purpose a standardized two-point-discriminator (PADGETT DeMayo Two-Point Discrimination Device, Used for Post hand surgery diagnostic. MFID: PM-855) is used
two point discrimination | 12 weeks postoperative
  For this purpose a standardized two-point-discriminator (PADGETT DeMayo Two-Point Discrimination Device, Used for Post hand surgery diagnostic. MFID: PM-855) is used
two point discrimination | 24 weeks postoperative
  For this purpose a standardized two-point-discriminator (PADGETT DeMayo Two-Point Discrimination Device, Used for Post hand surgery diagnostic. MFID: PM-855) is used

SECONDARY OUTCOMES:
Neuroma formation | 6 weeks postoperative
  * presence of Hofmann-Tinel sign
  * Allodynographia/Mapping (Semmes-Weinstein Monofilament (SWMF) assessment as described by Spicher et al. (17); Sammons Preston Rolyan) performed by a trained hand therapist
  * detection of a neuroma in ultrasound examination (measurement of three cross-section areas: proximal, distal and at the level of the neurorrhaphy) performed by a therefore certified hand surgeon (Philips iU22 Medical system or Philips 70 affiniti)
Grip strength | 12 weeks postoperative
  using a JAMAR dynamometer
Active range of motion | 6 weeks postoperative
  using a goniometer
Pain with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain | 6 weeks postoperative
  with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain
quickDASH score (Disabilities of the Shoulder, Arm and Hand) | preoperative
  a 11 item questionnaire: filled out by the patient
STI-Test: (Shape-Texture Identification test) | 12 weeks postoperative
  This test is a standardized outcome measure of sensory function of the median and ulnar nerves of the hand: max. score for completed test = 6 points, min. score = 0
Neuroma formation | 12 weeks postoperative
  * presence of Hofmann-Tinel sign
  * Allodynographia/Mapping (Semmes-Weinstein Monofilament (SWMF) assessment as described by Spicher et al. (17); Sammons Preston Rolyan) performed by a trained hand therapist
  * detection of a neuroma in ultrasound examination (measurement of three cross-section areas: proximal, distal and at the level of the neurorrhaphy) performed by a therefore certified hand surgeon (Philips iU22 Medical system or Philips 70 affiniti)
Neuroma formation | 24 weeks postoperative
  * presence of Hofmann-Tinel sign
  * Allodynographia/Mapping (Semmes-Weinstein Monofilament (SWMF) assessment as described by Spicher et al. (17); Sammons Preston Rolyan) performed by a trained hand therapist
  * detection of a neuroma in ultrasound examination (measurement of three cross-section areas: proximal, distal and at the level of the neurorrhaphy) performed by a therefore certified hand surgeon (Philips iU22 Medical system or Philips 70 affiniti)
Neuroma formation | 48 weeks postoperative
  * presence of Hofmann-Tinel sign
  * Allodynographia/Mapping (Semmes-Weinstein Monofilament (SWMF) assessment as described by Spicher et al. (17); Sammons Preston Rolyan) performed by a trained hand therapist
  * detection of a neuroma in ultrasound examination (measurement of three cross-section areas: proximal, distal and at the level of the neurorrhaphy) performed by a therefore certified hand surgeon (Philips iU22 Medical system or Philips 70 affiniti)
Grip strength | 24 weeks postoperative
  using a JAMAR dynamometer
Grip strength | 48 weeks postoperative
  using a JAMAR dynamometer
Active range of motion | 12 weeks postoperative
  using a goniometer
Active range of motion | 24 weeks postoperative
  using a goniometer
Active range of motion | 48 weeks postoperative
  using a goniometer
Pain with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain | 12 weeks postoperative
  with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain
Pain with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain | 24 weeks postoperative
  with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain
Pain with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain | 48 weeks postoperative
  with the Numeric Rating Scale (NRS): 0 indicating no and 10 indicating maximum pain
quickDASH score (Disabilities of the Shoulder, Arm and Hand) | 6 weeks postoperative
  a 11 item questionnaire: filled out by the patient
quickDASH score (Disabilities of the Shoulder, Arm and Hand) | 12 weeks postoperative
  a 11 item questionnaire: filled out by the patient
quickDASH score (Disabilities of the Shoulder, Arm and Hand) | 24 weeks postoperative
  a 11 item questionnaire: filled out by the patient
quickDASH score (Disabilities of the Shoulder, Arm and Hand) | 48 weeks postoperative
  a 11 item questionnaire: filled out by the patient
STI-Test: (Shape-Texture Identification test) | 24 weeks postoperative
  This test is a standardized outcome measure of sensory function of the median and ulnar nerves of the hand: max. score for completed test = 6 points, min. score = 0
STI-Test: (Shape-Texture Identification test) | 48 weeks postoperative
  This test is a standardized outcome measure of sensory function of the median and ulnar nerves of the hand: max. score for completed test = 6 points, min. score = 0

CONTACTS AND LOCATIONS:
Overall Officials: Esther Vögelin, Prof. Dr., Study Chair — Insel Gruppe AG, University of Bern
Locations (1):
- Insel Gruppe AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No